CLINICAL TRIAL: NCT06210789
Title: Periodontal Plastic Surgical Approaches to Correct Recession and Lack of Keratinized Tissue After Elimination of Localized Gingival Enlargements - a Case Series
Brief Title: Periodontal Plastic Reconstruction of Soft Tissue Dehiscences After the Removal of Localized Gingival Enlargements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Balint Molnar, Associate professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epulis
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Localized Gingival Enlargement; Epulides; Recurrence; Periodontal; Lesion
Keywords: Periodontal reconstructive surgery; Surgical excision; Surgical treatment; Localized Gingival Enlargement
MeSH Terms: conditions — Gingival Diseases; Recurrence

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgical treatment (Experimental): Surgical excision and periodontal reconstruction according to the remaining amount of keratinized gingiva
  Interventions: Procedure: Surgical excision

INTERVENTIONS:
Procedure: Surgical excision — Periodontal plastic reconstruction of the subsequent soft tissue dehiscence after the surgical excision of the localized gingival enlargement
  Other Names: periodontal plastic reconstruction

SUMMARY:
Non-inflammatory recessions and Miller class I-II-III. mucogingival defects after elimination of localized gingival enlargements are frequently encountered challenges in the daily practice. In Miller class II-III. recessions the lack of keratinized tissues often compromise the maintenance a proper oral hygiene, this can cause inflammation, which can result in further periodontal attachment loss. In the literature there are some approaches that aim at widening of keratinized tissues and root coverage at the same time, such as the subperiosteal envelope technique (SET) (Allen 1994) combined with a subepithelial connective tissue graft (SCTG) or a partially epithelialized connective tissue graft (PE-SCTG) (Stimmelmayr 2011). In the eradication of localized gingival enlargement postoperative complications following surgical removal, such as recurrence and subsequent gingival recessions as well as loss of keratinized tissues are commonly observed. Nevertheless, a state of the art comprehensive treatment approach has not been reported yet to overcome the above mentioned sequels. The aim of this study is to present a periodontal plastic surgical approach to definitively eliminate localized gingiva enlargements and to simultaneously correct consecutive Miller class I II-III. recessions, esthetic disturbances. (Ethical committee permission number: SE RKEB: 185/2020.)

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* systematically healthy patients
* localized gingival enlargement is present that involves maximum 3 teeth

Exclusion Criteria:

* pregnant women
* medication intake that can potentially affect the oral mucosa and its healing
* heavy smokers (>=15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 3 months, 6 months
  If there is recurrence after the proper elimination of the enlargement and the one-staged reconstruction

SECONDARY OUTCOMES:
Keratinized Gingiva Height | 1 month, 3 months, 6 months
  The height of the remaining keratinized gingiva
Gingival Recession | 1 month, 3 months, 6 months
  The subsequent gingiva recession that remains after the elimination of the enlargement and the reconstruction of the soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Bálint Molnár, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Faculty of Dentistry, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao N, Yesibulati Y, Xiayizhati P, He YN, Xia RH, Yan XZ. A large-cohort study of 2971 cases of epulis: focusing on risk factors associated with recurrence. BMC Oral Health. 2023 Apr 20;23(1):229. doi: 10.1186/s12903-023-02935-x. PMID 37081478
- See also: Institutional homepage — https://semmelweis.hu/parodontologia/en/